CLINICAL TRIAL: NCT03354507
Title: Use of Sodium Bicarbonate to Alkalinize Serum/Urine in Pediatric Patients Treated With Topiramate (Pilot Study)
Brief Title: Use of Sodium Bicarbonate in Patients Treated With Topiramate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster Children's Hospital (Other)
Responsible Party: Principal Investigator, Mandeep Sidhu, Resident Physician, McMaster Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1137
Record Dates: First submitted 2017-11-21; First posted 2017-11-28 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Epilepsy; Metabolic Acidosis; Tubular Acidosis; Renal
Keywords: topiramate; epilepsy; sodium bicarbonate; urine alkalinization
MeSH Terms: conditions — Epilepsy; Acidosis; Acidosis, Renal Tubular | interventions — Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium Bicarbonate (Experimental): Patients will receive sodium bicarbonate for 4 weeks, based on pre-calculated weight based doses. Patients are selected if they have metabolic acidosis at baseline.
  < 24 kg : 1/4 teaspoon bid. 24 - 42 kg : 1/2 teaspoon bid. > 42kg : 3/4 teaspoon bid.
  Interventions: Dietary Supplement: Sodium bicarbonate
- Control (No Intervention): Patients will not receive treatment if they do not have metabolic acidosis at baseline.

INTERVENTIONS:
Dietary Supplement: Sodium bicarbonate — Sodium bicarbonate. See arms.
  Arms: Sodium Bicarbonate

SUMMARY:
Effect of oral sodium bicarbonate therapy on renal tubular acidosis in epilepsy patients taking topiramate.

DETAILED DESCRIPTION:
Children on topiramate are at a risk of renal tubular acidosis and subsequent development of renal stones. Sodium bicarbonate has been shown to reduce renal tubular acidosis in other populations. To date, no data exist on the efficacy of correction of renal tubular acidosis in pediatric patients on topiramate. We are proposing to investigate the efficacy of 4 weeks of oral sodium bicarbonate therapy to reduce tubular acidosis in patients on topiramate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with epilepsy receiving oral topiramate for a minimum of 3 months

Exclusion Criteria:

* pre-existing renal impairments (ie nephropathy, primary nephritis)
* receiving other medications or diet therapies that may influence renal function or urine acidity/ citrate concentration

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Changes in measured urine parameters | Baseline, then at 4 weeks
  Spot urine sample will be tested for calcium, creatinine and citrate

SECONDARY OUTCOMES:
Changes in measured blood parameters. | Baseline, then at 4 weeks
  sodium, potassium, chloride, calcium, magnesium, phosphate, bicarbonate, alkaline phosphatase, urea, creatinine, venous blood gas
Changes in frequency of seizures. | Baseline, then at 4 weeks
  Changes in seizure entries in seizure diary

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ben-Menachem E, Sander JW, Stefan H, Schwalen S, Schauble B. Topiramate monotherapy in the treatment of newly or recently diagnosed epilepsy. Clin Ther. 2008 Jul;30(7):1180-95. doi: 10.1016/s0149-2918(08)80045-8. PMID 18691980
- [Background] Caudarella R, Vescini F. Urinary citrate and renal stone disease: the preventive role of alkali citrate treatment. Arch Ital Urol Androl. 2009 Sep;81(3):182-7. PMID 19911682
- [Background] Coe FL, Evan A, Worcester E. Kidney stone disease. J Clin Invest. 2005 Oct;115(10):2598-608. doi: 10.1172/JCI26662. PMID 16200192
- [Background] Dell'Orto VG, Belotti EA, Goeggel-Simonetti B, Simonetti GD, Ramelli GP, Bianchetti MG, Lava SA. Metabolic disturbances and renal stone promotion on treatment with topiramate: a systematic review. Br J Clin Pharmacol. 2014 Jun;77(6):958-64. doi: 10.1111/bcp.12283. PMID 24219102
- [Background] Hall PM. Nephrolithiasis: treatment, causes, and prevention. Cleve Clin J Med. 2009 Oct;76(10):583-91. doi: 10.3949/ccjm.76a.09043. PMID 19797458
- [Background] HANLEY T, PLATTS MM. Observations on the metabolic effects of the carbonic anhydrase inhibitor diamox: mode and rate of recovery from the drug's action. J Clin Invest. 1956 Jan;35(1):20-30. doi: 10.1172/JCI103248. No abstract available. PMID 13278397
- [Background] Mirza N, Marson AG, Pirmohamed M. Effect of topiramate on acid-base balance: extent, mechanism and effects. Br J Clin Pharmacol. 2009 Nov;68(5):655-61. doi: 10.1111/j.1365-2125.2009.03521.x. PMID 19916989
- [Background] Moher D, Liberati A, Tetzlaff J, Altman DG; PRISMA Group. Preferred reporting items for systematic reviews and meta-analyses: the PRISMA statement. Ann Intern Med. 2009 Aug 18;151(4):264-9, W64. doi: 10.7326/0003-4819-151-4-200908180-00135. Epub 2009 Jul 20. No abstract available. PMID 19622511
- [Background] Silberstein SD, Ben-Menachem E, Shank RP, Wiegand F. Topiramate monotherapy in epilepsy and migraine prevention. Clin Ther. 2005 Feb;27(2):154-65. doi: 10.1016/j.clinthera.2005.02.013. PMID 15811478
- [Background] Vega D, Maalouf NM, Sakhaee K. Increased propensity for calcium phosphate kidney stones with topiramate use. Expert Opin Drug Saf. 2007 Sep;6(5):547-57. doi: 10.1517/14740338.6.5.547. PMID 17877442
- [Background] Wile D. Diuretics: a review. Ann Clin Biochem. 2012 Sep;49(Pt 5):419-31. doi: 10.1258/acb.2011.011281. Epub 2012 Jul 10. PMID 22783025